CLINICAL TRIAL: NCT06599372
Title: Treatment of Resistant Auditory Hallucinations in Schizophrenia by Repetitive Transcranial Magnetic Stimulation. Naturalistic Study
Brief Title: Evaluation of the Efficacy of Transcranial Magnetic Stimulation on Resistant Auditory Hallucinations in Schizophrenia
Acronym: HRRENAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dominique JANUEL (Other)
Responsible Party: Sponsor-Investigator, Dominique JANUEL, Head of clinical research unit, Centre hospitalier de Ville-Evrard, France
Organization: Centre hospitalier de Ville-Evrard, France (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-A02698-33
Record Dates: First submitted 2024-07-24; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Schizophrenia; Transcranial Magnetic Stimulation; Hallucinations, Verbal Auditory
Keywords: hallucinations; resistant auditory hallucinations; schizophrenia; TMS; Transcranial magnetic stimulation; TBS; Theta burst stimulation; a improvement; real-life conditions
MeSH Terms: conditions — Schizophrenia; Hallucinations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The rTMS method (Other): The treatment lasts 2 weeks with 20 rTMS sessions at a rate of 2 sessions per day. Each session lasts 20 minutes with a one hour break between sessions. The application of rTMS will be done on the left temporo-parietal junction.
  Interventions: Other: The rTMS method
- The cTBS method (Other): The treatment lasts 15 days with 45 sessions of cTBS at a rate of 3 sessions per day. The session lasts 40 seconds and consists of 3 pulses at 50Hz repeated every 200 milliseconds (5Hz) to reach a total of 600 pulses, with a 15 minute break between sessions. The application of cTBS will be performed on the left temporo-parietal junction.
  Interventions: Other: The cTBS method

INTERVENTIONS:
Other: The rTMS method — The patient receives treatment under naturalistic conditions in routine practice.
  Arms: The rTMS method
Other: The cTBS method — The patient receives the treatment under naturalistic conditions in routine practice.
  Arms: The cTBS method

SUMMARY:
This open naturalistic study aims to evaluate the efficacy of rTMS in routine practice on auditory resistant hallucinations (AHR) of patients with schizophrenia. To this end, two stimulation methods will be offered to patients: the rTMS stimulation method and the cTBS stimulation method.We principally use the AHRS scale to evaluate the effectiveness of rTMS on RAH in patients with schizophrenia. Our main hypothesis is that rTMS used under naturalistic conditions, in addition to antipsychotics, would allow a relative improvement of resistant auditory hallucinations assessed by the AHRS scale between baseline and end of treatment in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient diagnosed with schizophrenia according to DSM-V criteria (Diagnostic and Statistical Manual of Mental Disorder V5, 2013)
* Presence of auditory hallucinations: Resistant auditory hallucinations: resistance to treatment with 2 different well-conducted antipsychotics.
* Patient agreeing to participate in the study and having signed an informed consent
* Patient with French language skills
* Affiliation to a social security system
* Women of childbearing age must be on contraception and have a negative pregnancy test (βHCG)

Exclusion Criteria:

* Have a contraindication to MST: intracranial foreign body, unstabilized epilepsy, cochlear implant
* Presence of an unstabilized medical condition
* Pregnant woman (Women of childbearing age without effective contraception)
* Current or less than one month old engagement in another research protocol
* A person who is subject to a safeguard of justice measure
* An adult under curatorship
* Minor patients with mental health problems
* Pregnant or breastfeeding women
* A person in a social fragility (Persons deprived of liberty by a judicial or administrative decision, hospitalized persons)
* Persons incapable or unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The evolution will be evaluated mainly with the AHRS (Auditory Hallucinations Rating Scale) | Baseline and at the end of the treatment, also at 1 month and 3 months after the end of the treatment
  Refer to the definition of AHRS above (in Primary Outcome Measure)

SECONDARY OUTCOMES:
Response rate: a response is defined as a decrease greater than or equal to 30% of total AHRS score from baseline to end of treatment. | Baseline and at the end of the treatment
  Refer to the definition of AHRS above
Rate of patients with an end-of-treatment score < 3 on the Positive And Negative Syndrome Scale (PANSS) "Hallucinatory Behavior" item | Baseline and at the end of the treatment
  The PANSS is a 30 items scale rated from 1 (absent) to 7 (extreme), that assesses psychopathological symptoms observed in patients with psychotic states, particularly schizophrenia.
Cognitive symptoms: Montreal Cognitive Assessment (MOCA), Stroop | Baseline and 1 month after the end of treatment
  The MoCA scale is the most sensitive rapid assessment test and provides the broadest evaluation of cognitive functions (attention, concentration, executive functions, memory, language, visualconstructive abilities, abstraction, calculation, orientation). It tends to replace the MMSE in clinical practice. A score < 26 (25 if cultural level < 3 = primary diploma = CEP) is considered abnormal. The Stroop scale evaluates the capacity for attention and inhibition; thus, it allows to measure the level of interference generated by the automatisms in the accomplishment of a task. The result of the test allows us to see if the person is correctly inhibiting the response (values greater than 0, positive) or if there are significant interference problems (if it is a negative value).
Addictive attitudes: number of cigarettes/d (tobacco), The Cannabis Abuse Screening Test (CAST), Marijuana Craving Questionnaire (MCQ) | Baseline and at the end of the treatment
  The CAST is a 6-item scale for identifying problematic cannabis use. Each of these items describes use behaviors or problems encountered with cannabis use. The CAST score determines the patient's level of dependence. A score of 1 or less means low risk. A score of 2 means moderate risk. A score of 3 or higher means high risk. The MCQ self-report scale is a questionnaire on marijuana craving. It consists of four constructs or factors that characterize cannabis craving: compulsivity, emotionality, expectancy and determination. A separate score is calculated for each factor. The MCQ can be used to measure cue-induced craving in a research setting or natural craving in cannabis-dependent individuals presenting for treatment.
Mood: Calgary Depression Scale for Schizophrenia (CDSS) | Baseline and the end of the treatment
  The CDSS, is designed to assess depression in people with schizophrenia. It takes into account negative symptomatology and possible extrapyramidal effects of neuroleptics. The questionnaire consists of 9 items covering the last 2 weeks. Each item is evaluated on a 4 points Likert scale ranging from : "Absent" (0) to "Severe" (3). The total score is obtained by adding the items and gives a score out of 27.
Quality of life: The Subjective Quality of Life Scale (S-QoL) | Baseline and end of treatment, also at 1 month and 3 months after the end of the treatment
  The SQoL questionnaire is a self-administered quality of life scale that assesses quality of life in people with schizophrenia from the patient's perspective. The questionnaire has 18 items, each item is rated on a 4 points Likert scale ranging from: "Much less" to "More than desired". Scores range from 0 to 100; higher scores represent better quality of life.
Clinical Global Impressions (CGI) Scale | Baseline and end of treatment, also at 1 month and 3 months after the end of the treatment
  Clinical Global Impression (CGI) scales are measures of symptom severity, response to treatment, and treatment effectiveness in treatment studies of patients with mental disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique JANUEL, Study Director — Clinical research unit, EPS Ville Evrard; Noomane BOUAZIZ, Principal Investigator — Clinical research unit, EPS Ville Evrard
Locations (1):
- Etablissement Public de Santé de Ville-Evrard, Neuilly-sur-Marne, France